CLINICAL TRIAL: NCT07230912
Title: Impact of Comorbidities, Some Biomarkers, Micro RNA in Childhood Asthma Phenotypes, Severity and Response to Therapy
Brief Title: Impact of Comorbidities, Some Biomarkers, Micro RNA in Childhood Asthma Phenotypes
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aghapy Gamal Zahy Shafik, Assistant lecteurer of pediatrics, Assiut University
Other Study IDs: bronchial asthma in children
Record Dates: First submitted 2025-10-02; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- comparing the mean of FEV1 between two independent groups(comorbidity in bronchial asthma )
  Interventions: Drug: Short Acting Beta 2 Agonist

INTERVENTIONS:
Drug: Short Acting Beta 2 Agonist — short acting drug

SUMMARY:
* Assess response to treatment in children with bronchial asthma attending Assiut university children hospital.
* Role of comorbidities in controlling symptoms of bronchial asthma.
* Evaluate the role of the soluable interleukin 5 receptor, I C-telopeptide of type I collagen (ICTP), miR-223-3p and miR-191-5p in bronchial asthma.

DETAILED DESCRIPTION:
Asthma is a heterogenous disease usually characterized by chronic air way inflammation. It is defined by the history of respiratory symptoms such as wheeze, shortness of breath, chest tightness and cough. Asthma affects approximately 300 million people around the world causing about 1,000 deaths per day.

The overall prevalence of asthma among children and adolscents in Eastern Mediterranean Regional Office (EMRO) countries was 10.61%, Among the countries studied, Qatar exhibited the highest prevalence at 16.69%, Egypt (8.85%), Adolescents showed a slightly higher prevalence of asthma at 10.10% compared to children at 9.70%. Boys exhibited a higher prevalence at 11.48% compared to girls at 9.75%. Urban areas demonstrated a higher prevalence at 11.27% than rural areas at 8.29%.

In recent decades, both asthma prevalence and incidence have been increasing worldwide, not only due to the genetic background, but mainly to the effect of a wide number of environmental risk factors, many of which included under the umbrella of "modern lifestyle". However, the worldwide economic globalization could also have contributed to a significant increase in the asthma burden, even in developing countries that presented a low disease prevalence in the recent past.

Severe asthma is an important health burden as children with severe asthma are prone to medication related side effects, life threatening exacerbations, and impaired quality of life. Progressive air flow limitation is also a feature of severe asthma. Most importantly, poor asthma control leads to poor quality of life in children and caregivers.

Comorbidities such as cardiovascular, metabolic, endocrine, respiratory, and psychiatric diseases are prevalent in asthma, owing to chronic inflammation, systemic corticosteroid use, reduced physical activity, and poor sleep.

These comorbidities may obscure asthma diagnosis by mimicking the symptoms of the disease and can influence management, owing to the effects of the treatments of the comorbidities on asthma or of asthma therapy on the comorbid conditions.

Comorbidities with a major impact are rhinitis (particularly in its allergic form), which causes inflammation of the upper airways and can contribute to exacerbate asthma, gastroesophageal reflux (GERD), which may aggravate airway inflammation, obesity, which not only affects respiratory mechanics but induces a systemic proinflammatory status; and, bronchiectasis, which exposes the patient to an increased risk for exacerbations owing to pulmonary infections.

In addition to these, environmental allergen control is an important contributor to poor asthma control. Ongoing allergen or irritant exposure at home or school will end up with difficult to treat asthma.

Addressing comorbidities of asthma is very important for better asthma control. increased BMI, GERD, sinusitis are significantly associated with exacerbation frequency. Evaluation for those disorders should be considered.

Identifying how comorbidities affect disease control in different groups of patients will allow a more personalized approach, focusing on the treatment of individual characteristics and avoiding escalation to maximal therapy.

Asthma is a heterogenous disease in which age of onset has emerged as an important determinant of different phenotypes. Childhood-onset asthma is approximately 70% atopic, with T-helper-2 (Th2) type of airway inflammation, corticosteroid treatment responsiveness, and a good prognosis.

Th2-type cytokines, such as interleukin 4 (IL-4), IL-5, and IL-13, are thought to drive the disease pathology in patients with asthma and play a role in driving many of the hallmarks of allergic inflammation. IL-5 is the critical molecular switch for developing, migrating, and recruiting eosinophils to the lung during allergic inflammation. IL-5 exerts its biological actions via stimulation of the IL-5 receptor expressed by eosinophils, and to a lesser extent, also by basophils.

A range of biomarkers have been identified for the high TH2 asthma, but biomarkers for non-TH2 asthma endotype, also known as the non-eosinophilic asthma endotype, are lacking. However, sputum neutrophils, blood neutrophils, and IL-17 have been proposed as markers for the noneosinophilic endotype.

During airway tissue remodeling, subepithelial fibrosis leads to an altered extracellular matrix (ECM) content, contributing to asthma's pathogenesis . The existence of subepithelial fibrosis in asthmatic airways suggests an imbalance between matrix metalloproteinases (MMP) and their inhibitors.

Type I collagen is one of the most abundant collagens in the healthy lung, providing a structural framework for the airway wall. Type I collagen plays a significant constitute in subepithelial fibrosis in asthmatic airways.

MicroRNAs (miRNAs) are small, non-coding RNA molecules with a length of 21-25 nucleotides. MiRNAs can control gene expression by targeting specific mRNAs for degradation or translational repression. MiRNAs bind to a specific sequence at the 3'UTR of the target messenger RNA (mRNA). The complementary sequences between miRNA and mRNA are usually not fully overlapping, implicating that each miRNA can regulate hundreds of target genes and that several miRNAs can target the same mRNAs.

MiR-223 has a crucial role in innate immunity, myeloid cell differentiation, and cell homeostasis and has several targets that are involved in pathways implicated in the pathogenesis of both asthma and COPD. Finally, miR-223 is easily detectable in multiple human samples (e.g., sputum, bronchial biopsies, and blood) and could therefore serve as a potential biomarker.

levels of miR-191-5p was upregulated in extracellular vehicles (EVs) derived from individuals with asthma, indicating a possible association with both lung function deterioration and inflammation . EVs, as intercellular communication and delivery systems, can play key roles in different pathological and physiological body functions. Research has indicated that EVs containing miR-191-5p may promote inflammatory responses, aggravating asthma symptoms by activating the NF-κB pathway.

Effective asthma management involves a holistic approach addressing both pharmacological and non-pharmacological management, as well as education and self-management aspects. Working in partnership with children and families is key in promoting good outcomes. Education on how to take treatment effectively, trigger avoidance, modifiable risk factors and actions to take during acute attacks via personalised asthma action plans is essential.

All children aged 5 years or younger with asthma or suspected asthma should be provided with inhaled SABA for relief of symptoms. Regular daily low dose ICS is recommended as initial treatment to control asthma in children aged 5 years or For children 6-11 years with asthma symptoms that are well controlled on low dose ICS or who are using SABA alone and have symptoms less than twice aweek, the recommended treatment is taking ICS whenever SABA is taken.

The use of these inhalers have been shown to reduce the risk of asthma attacks and emergency department (ED) admissions, improve lung function and decrease the need for reliever therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years diagnosed asthma, inpatient or attending pediatric outpatient clinic of Assiut university children hospital.

Exclusion Criteria:

* - Chronic respiratory illness other than asthma (e.g., bronchiectasis, CF)
* Known immunodeficiency or systemic illness
* patients with skeletal deformities
* patients suspected inborn errors of metabolism

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Data Collection Tools:
  History
  * Personal history
  * A detailed history including the outline of respiratory symptoms, triggers for cough, wheeze, shortness of breath
  * Asthma history (duration, triggers, control status)
  * Therapeutic history (medications used during previous 12 months) History suggestive of GERD as: heart burn, regurgitation, vomiting
  * Past history of other allergic diseases as: Allergic rhinitis ,urtcaria and food allergy
  * positive family history of asthma and other allergic diseases Complete physical examination
  * BMI to assess obesity
  * Chest examination
  Investigations:
  * CBC (neutrophils-esinophils)
  * Inflammatory markers (ESR-CRP)
  * Total IgE
  * lipid profile
  * The soluable interleukin 5 receptor 1
  * I C-telopeptide of type I collagen (ICTP)
  * miR-223-3p
  * miR-191-5p chest xray Pulmonary function test (spirometry) follow up patients as regards asthma control,exacerbation in one year
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
-proportion of participants achieving clinical treatment response (forced expiratory volume in one second (FEV1) increase >12% from baseline). -association between baseline circulating micro RNA (miR-223-3p- miR-191-5p) and clinical treatment response. | one year
  * number and percentage of children showing improvment in lung function defined as an increase in forced expiratory volume in one second >12 from baseline measured by standardized spirometry (pre and post bronchodilator) at one year.
  * correlation and between- group differences in baseline serum micoRNA levels (miR-223-3p- miR-191-5p) comparing responders vs non-responders in 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mahrous El Tallawy, professor of pediatrics, Study Chair — Assiut university children hospital; Yasser Gamal Abdel-Rahman, Assistant Professor, Principal Investigator — Assiut university children hospital; Ahmed Zohri Yasin, Lecturer of Pediatrics, Study Director — Assiut university children hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roffel MP, Bracke KR, Heijink IH, Maes T. miR-223: A Key Regulator in the Innate Immune Response in Asthma and COPD. Front Med (Lausanne). 2020 May 19;7:196. doi: 10.3389/fmed.2020.00196. eCollection 2020. PMID 32509795
- [Result] Vafadar A, Alashti SK, Khazayel S, Babadi S, Eghtesadi M, Younesi M, Savardashtaki A, Negahdaripour M. Meta-analysis of microarray data to identify potential signature genes and MiRNAs associated with the pathogenesis of asthma. J Transl Med. 2025 Jul 15;23(1):796. doi: 10.1186/s12967-025-06646-5. PMID 40665411
- [Result] Martin J, Townshend J, Brodlie M. Diagnosis and management of asthma in children. BMJ Paediatr Open. 2022 Apr;6(1):e001277. doi: 10.1136/bmjpo-2021-001277. PMID 35648804
- [Result] Sobieraj DM, Weeda ER, Nguyen E, Coleman CI, White CM, Lazarus SC, Blake KV, Lang JE, Baker WL. Association of Inhaled Corticosteroids and Long-Acting beta-Agonists as Controller and Quick Relief Therapy With Exacerbations and Symptom Control in Persistent Asthma: A Systematic Review and Meta-analysis. JAMA. 2018 Apr 10;319(14):1485-1496. doi: 10.1001/jama.2018.2769. PMID 29554195
- [Result] Taherian MR, Fatemian F, Halimi A, Soleimani Y, Jorjani G, Nozari P, Mosavi Jarrahi A, Nazari SSH, Al-Yateem N, Al-Marzouqi A, Humid A, Rahman SA. Prevalence of asthma among children and adolescents in WHO's Eastern Mediterranean Region: a meta-analysis of over 0.5 million participants. BMC Public Health. 2024 Aug 7;24(1):2148. doi: 10.1186/s12889-024-18716-2. PMID 39112964